CLINICAL TRIAL: NCT01087814
Title: Effect of Encapsulation Upon Efavirenz Pharmacokinetics
Brief Title: Sustiva Levels With Use of a Gel Capsule
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 0910M73917
Record Dates: First submitted 2010-03-15; First posted 2010-03-16 (Estimated); Results first posted 2014-09-12 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-01

CONDITIONS: HIV; HIV Infections
Keywords: efavirenz; Sustiva; pharmacokinetics
MeSH Terms: conditions — HIV Infections | interventions — efavirenz

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- efavirenz (Active Comparator)
  Interventions: Drug: Efavirenz
- over-encapsulated efavirenz (Experimental)
  Interventions: Drug: Over-encapsulated efavirenz

INTERVENTIONS:
Drug: Efavirenz — Subject will take efavirenz for 5 days.
  Other Names: Sustiva
  Arms: efavirenz
Drug: Over-encapsulated efavirenz — Subject will take efavirenz that has been over-encapsulated with a gel capsule for 5 days.
  Other Names: Over-encapsulated Sustiva
  Arms: over-encapsulated efavirenz

SUMMARY:
We are studying if putting a gel capsule over a standard HIV drug changes the ability of the body to absorb the drug. This is important because we want to be able to study new HIV drugs against the most common drugs used today and the most common is Sustiva, which is also called efavirenz. We will give you Sustiva every day for 5 days and draw blood to see how much is absorbed. Then we will give you Sustiva that has a gel capsule over it for 5 days and we will draw blood to see how much is absorbed.

ELIGIBILITY:
Inclusion Criteria:

* HIV-negative, proven by ELISA
* Age: ≥ 18 years old

Exclusion Criteria:

* Psychiatric or psychological illness that would make adherence to protocol procedures unlikely.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-02; Primary Completion 2010-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy W Schacker, M.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Efavirenz First, Then Over-encapsulated Efavirenz: This arm received efavirenz for five days, then over-encapsulated efavirenz for five days.
- Over-encapsulated Efavirenz First, Then Efavirenz: This arm received over-encapsulated efavirenz for five days, then efavirenz for five days.
Period: First Intervention (5 Days)
Arm/Group | Efavirenz First, Then Over-encapsulated Efavirenz | Over-encapsulated Efavirenz First, Then Efavirenz
Started | 8 | 7
Completed | 5 | 6
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 3 | 1
Period: Second Intervention (5 Days)
Arm/Group | Efavirenz First, Then Over-encapsulated Efavirenz | Over-encapsulated Efavirenz First, Then Efavirenz
Started | 5 | 6
Completed | 4 | 6
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Efavirenz: Both arms received both versions of the drug during the course of the study.
- Over-encapsulated Efavirenz: Both arms received both versions of the drug over the course of the study.
- Total: Total of all reporting groups
Arm/Group | Efavirenz | Over-encapsulated Efavirenz | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 7 | 15
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.125 (8.45893) | 25.875 (2.53194) | 26 (6.03324)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Serum Levels of Efavirenz
Description: Serum levels of efavirenz were measured on the fifth day of taking efavirenz (tablet) and the fifth day of taking an overencapsulated efavirenz.
Time Frame: 5th day of taking drug
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Efavirenz (Tablet): All subjects took efavirenz.
- Over-encapsulated Efavirenz: All subjects took over-encapsulated efavirenz.
Arm/Group | Efavirenz (Tablet) | Over-encapsulated Efavirenz
Number analyzed (Participants) | 10 | 10
ng/mL | 5151.11 (765.67) | 4965.08 (1285.48)

ADVERSE EVENTS:
Arm/Group | Efavirenz | Over-encapsulated Efavirenz
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 0/8 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No